CLINICAL TRIAL: NCT06012123
Title: COMBINATION OF BEGRAFT AND SOLARIS STENTGRAFTS FOR THE COVERED ENDOVASCULAR RECONSTRUCTION OF AORTIC BIFURCATION (BS-CERAB) TECHNIQUE
Brief Title: BS-CERAB TECHNIQUE
Acronym: BS-CERAB
Status: Completed | Type: Observational
Sponsor: Vascular Investigation Network Spanish Society for Angiology and Vascular Surgery (Network)
Responsible Party: Sponsor
Other Study IDs: PI23-0005
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Aortoiliac Occlusive Disease; Stent Complication; Vascular Device Occlusion; Iliac Artery Stenosis
MeSH Terms: interventions — Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Aortoiliac angioplasty and stenting — Covered endovascular reconstruction of aortic bifurcation (CERAB) in patient with aorto-iliac occlusive disease

SUMMARY:
The covered endovascular reconstruction of aortic bifurcation (CERAB) technique was described l in 2013 to reconstruct the aortic bifurcation in a more anatomical and physiological way. With the use of this technique, a covered stent is expanded 15 to 20 mm above the aortic bifurcation and this stent is proximally adapted to the aortic wall with a larger balloon, thereby creating a cone-shaped stent. Two iliac covered stents are then placed in the distal conic segment and simultaneously inflated, making a tight connection with the aortic stent, as if they were molded together, thus simulating a new bifurcation. This minimal invasive endovascular technique using covered stents, was developed in order to optimize endovascular mimicking the anatomical configuration of the aortic bifurcation and in an attempt to overcome the disadvantages of kissing stents influenced by geometric factors such as radial mismatch, protrusion mismatch and stent conformation. The use of BeGraft (balloon-expandalbe covered stent) and Solaris (self-expandable covered stent) fro this technique is revised.

DETAILED DESCRIPTION:
The covered endovascular reconstruction of aortic bifurcation (CERAB) technique was described l in 2013 to reconstruct the aortic bifurcation in a more anatomical and physiological way.

With the use of this technique, a covered stent is expanded 15 to 20 mm above the aortic bifurcation and this stent is proximally adapted to the aortic wall with a larger balloon, thereby creating a cone-shaped stent. Two iliac covered stents are then placed in the distal conic segment and simultaneously inflated, making a tight connection with the aortic stent, as if they were molded together, thus simulating a new bifurcation.

This minimal invasive endovascular technique using covered stents, was developed in order to optimize endovascular mimicking the anatomical configuration of the aortic bifurcation and in an attempt to overcome the disadvantages of kissing stents influenced by geometric factors such as radial mismatch, protrusion mismatch and stent conformation.

The use of BeGraft (balloon-expandalbe covered stent) and Solaris (self-expandable covered stent) fro this technique is revised.

A retrospective study included patients that underwent endovascular treatment of atherosclerotic steno-occlusive aorto-iliac lesions between January 2020 and June 2023. The study, which received no financial support from industry, was performed in agreement with the Declaration of Helsinki and was approved by our institutional review boards. In accordance with institutional and local regulatory policies, this retrospective review of de-identified procedural and follow-up data was exempt from informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lifestyle-limiting intermittent claudication, ischemic rest pain, ischemic ulcers or gangrene (Rutherford class 3 to 6) who presented steno-occlusive disease of the aortic bifurcation undergoing endovascular treatment by CERAB and PTA/covered stenting of iliac arteries

Exclusion Criteria:

* Patients who could not receive antiplatelet or anticoagulation therapies.
* Patients with concomitant aneurysm of the aorta, acute thrombus, unsalvageable limb or very limited life-expectancy.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that underwent endovascular treatment of atherosclerotic steno-occlusive aorto-iliac lesions between January 2020 and June 2023.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Primary patency | 12 months
  Absence of binary restenosis or reocclusion on duplex ultrasound examination without repeat target lesion interventions

SECONDARY OUTCOMES:
Primary-assisted patency | 12 months
  Patent aoto-iliac segment that underwent further intervention within the inflow, treated vessel segment, or outflow of the treated vessel segment to improve patency
Secondary patency | 12 months
  Requiring a secondary intervention to restore patency after occlusion of the treated segment. Secondary interventions include PTA, drug-eluting balloon PTA (DEB-PTA), additional stent placement or surgical bypass based on clinical deterioration.
Mortality | 12 months
Amputation rate | 12 months
  Major and minor amputation rate
Clinical status | 12 months
  Rutherford scale
ABI measurements | 12 months
  Ankle-Brachial index

CONTACTS AND LOCATIONS:
Locations (1):
- Valladolid Univeristy Hospital, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No
Investigation completion in 6 months, and publication in recognized clinical Journal